CLINICAL TRIAL: NCT01892449
Title: Comparison of Different Inspiratory to Expiratory Ratios on Respiratory Mechanics and Oxygenation in Robot-assisted Laparoscopic Radical Prostatectomy With Steep Trendelenburg Position and Pneumoperitoneum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2013-0287
Record Dates: First submitted 2013-06-30; First posted 2013-07-04 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: General Anesthesia Using Endotracheal Intubation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prolonged I:E ratio (1:1) group (Experimental)
  Interventions: Other: prolonged inspiratory to expiratory (I:E) ratio (1:1)
- conventional I:E ratio (1:2) group (Active Comparator)
  Interventions: Other: conventional I:E ratio (1:2)

INTERVENTIONS:
Other: prolonged inspiratory to expiratory (I:E) ratio (1:1) — 80 patients are randomly allocated into two groups : prolonged I:E ratio (1:1) (n=40) and conventional I:E ratio (1:2) group (n=40). In the prolonged I:E ratio (1:1), mechanical ventilation is maintained with during I:E ratio 1:1 during steep trendelenburg with pneumoperitoneum.
  Arms: prolonged I:E ratio (1:1) group
Other: conventional I:E ratio (1:2) — 80 patients are randomly allocated into two groups : prolonged I:E ratio (1:1) (n=40) and conventional I:E ratio (1:2) group (n=40). In the conventional I:E ratio (1:2) group (n=40), mechanical ventilation is maintained with during I:E ratio 1:2 during steep trendelenburg with pneumoperitoneum.
  Arms: conventional I:E ratio (1:2) group

SUMMARY:
The steep trendelenburg position and pneumoperitoneum during laparoscopic surgery have the potential to cause an adverse effects on respiratory mechanics and gas exchange. Previous studies have proposed that a prolonged I:E ratio ventilation improved respiratory mechanics and gas exchange. Therefore, the aim of this study is to evaluate whether a prolonged I:E ratio ventilation improves gas exchange and respiratory mechanics in patients undergoing robot-assisted laparoscopic radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patients (20-90 years of age) scheduled for elective robot-assisted laparoscopic radical prostatectomy undergoing general anesthesia

Exclusion Criteria:

* Patients with an abnormal airway anatomy, reactive airway diseases, chronic respiratory diseases, a history of coronary artery diseases, or heart failure
* BMI > 30 kg/m 2

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The peak inspiratory pressure | before 10 minutes after anesthesia induction, 30 and 60 minutes after steep trendelenburg position and pneumoperitoneum, and 10 minutes after supine position and CO2 desufflation
  The peak inspiratory pressure during mechanical ventilation with endotracheal intubation under general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Anesthesia and Pain Research Institute Yonsei University, Seoul, South Korea

REFERENCES:
- [Background] Al-Shaikh B, George William M, Van Zundert AA. Using atmospheric pressure to inflate the cuff of the Portex Laryngeal Mask. Anaesthesia. 2005 Mar;60(3):296-7. doi: 10.1111/j.1365-2044.2005.04135.x. No abstract available. PMID 15710025
- [Derived] Kim MS, Kim NY, Lee KY, Choi YD, Hong JH, Bai SJ. The impact of two different inspiratory to expiratory ratios (1:1 and 1:2) on respiratory mechanics and oxygenation during volume-controlled ventilation in robot-assisted laparoscopic radical prostatectomy: a randomized controlled trial. Can J Anaesth. 2015 Sep;62(9):979-87. doi: 10.1007/s12630-015-0383-2. Epub 2015 Apr 14. PMID 25869025